CLINICAL TRIAL: NCT02404233
Title: A Phase IV 48 Week, Open Label, Pilot Study of Darunavir Boosted by Cobicistat in Combination With Rilpivirine to Treat HIV+ Naïve Subjects (PREZENT)
Brief Title: Open Label, Pilot Study of Darunavir Boosted by Cobicistat in Combination With Rilpivirine to Treat HIV+ Naïve Subjects
Acronym: PREZENT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Therapeutic Concepts (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC278HIV4003
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: HIV Positive
MeSH Terms: conditions — HIV Seropositivity | interventions — cobicistat mixture with darunavir; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Darunavir/ cobicistat and Rilpivirine (Experimental): Single arm study:
  Darunavir/ cobicistat 800/ 150 mg tablet once daily taken with food Rilpivirine tablet 25 mg once daily taken with food
  Interventions: Drug: darunavir/cobicistat; Drug: rilpivirine

INTERVENTIONS:
Drug: darunavir/cobicistat — Darunavir/ cobicistat 800/ 150 mg tablet once daily taken with food
  Other Names: PREZCOBIX™ ; EDURANT®
Drug: rilpivirine — Rilpivirine tablet 25 mg once daily taken with food

SUMMARY:
Current HIV treatment guidelines recommend the use of triple-drug therapy (two nucleoside reverse transcriptase inhibitors and either a protease inhibitor, non-nucleoside reverse transcriptase inhibitor, or an integrase inhibitor) for the treatment of antiretroviral (ARV)-naïve patients. With the introduction of highly active antiretroviral therapy (HAART), patients with HIV are living much longer. With the increasing lifespan of persons with HIV, long-term complications from therapy as well as the occurrence of co-morbidities with aging have prompted HCPs to re-think the current treatment paradigm and consider novel combinations of ARVs. All of the currently approved HIV antiretrovirals have been implicated in causing long-term toxicities; however the greatest body of evidence for long-term metabolic effects has implicated the nucleoside reverse transcriptase (NRTI) class. By utilizing a non-NRTI treatment regimen, it is hypothesized that many of these long-term metabolic effects (renal toxicity, bone loss, body fat changes) can be delayed or avoided altogether. The clinical data on novel combinations is currently limited but rapidly growing and has included several combinations that have utilized darunavir. This study will be the first of its kind using the unique combination of darunavir/cobicistat and rilpivirine. Currently, this drug combination is not a recommended option for first time treatment of HIV

DETAILED DESCRIPTION:
This is a Phase IV, 48-week, open-label, pilot study in 30 ARV-naïve patients examining the safety, viral response, and tolerability of darunavir/cobicistat in combination with rilpivirine once daily for the treatment of HIV in treatment-naïve patients.

Thirty subjects meeting the inclusion criteria for study will be selected at a single site. All 30 subjects will receive darunavir/cobicistat 800/150mg in combination with rilpivirine 25 mg once daily at study onset and will be followed for 48 weeks after starting study medications. Virologic failure will be defined as failure to achieve HIV-1 RNA <50 copies/mL by week 24 of therapy, or in patients with baseline HIV-1 RNA >100,000 copies/mL, failure to achieve 1 log10 reduction in HIV-1 RNA by week 24. Confirmed virologic failure will be defined as two consecutive HIV RNA levels ≥50 copies/mL after suppression to <50 copies/mL for two consecutive measurements. Patients with confirmed virologic failure will be discontinued from the study and switched to a new antiretroviral treatment regimen.

Patients who have decided to initiate treatment after consultation with their physician and after careful review of the Department of Health and Human Services (DHHS) guidelines for treatment will be considered for enrollment as research subjects. Individuals considered for enrollment providing informed consent (See Appendix A) will be screened and, if eligible, enrolled in the study. Adherence to study regimen and symptoms of hypersensitivity reactions will be monitored by self-report at each study visit. Adherence will be assessed using the standard ACTG Adherence Questionnaire II (See Appendix B), either over the telephone or during a clinic visit. Those patients reporting problems with adherence will be counseled and monitored closely every 4 weeks at clinic visits with phone consultation bi-weekly until adherence improves. If despite counseling, adherence is not maintained, patients will be discontinued from the study due to increased risk of drug resistance. AEs will be monitored closely to determine if appropriate management affects tolerability and adherence, i.e., prescribing anti-emetic or anti-diarrhea medications for nausea and diarrhea, respectively. Patients will be counseled on the importance of adherence at every study visit.

Hematology, blood chemistry, liver function tests, virologic and immunologic measurements will be obtained at baseline (week 0), weeks 4, 12, 24, 36, and 48. In addition to blood chemistry evaluations, fasting blood samples will be obtained at baseline and weeks 24 and 48 for triglycerides, total cholesterol, direct HDL cholesterol and LDL cholesterol. Pancreatic amylase and serum lipase levels will be determined if serum amylase results are >2x ULN (see Section 5.4.2 Laboratory Evaluations).

In a subset of 12 subjects at their baseline and with at least 24 weeks exposure to darunavir and rilpivirine a lumbar puncture will be performed to obtain a sample of CSF for viral load, cell count and darunavir and rilpivirine concentration.

Adherence counseling will be performed after each HIV-1 RNA measurement of >400 copies/mL. New combination therapy for HIV will be initiated upon evidence of developing resistance in the face of virologic failure.

Samples for flow cytometry (including but not limited to absolute and percent CD4+ and CD8+ cell counts) and HIV RNA levels will be obtained at each study visit. The Roche Amplicor 1.5v (LOQ= 50 copies/mL) will be used until the patient has achieved an HIV RNA level < 50 copies/mL at which time the HIV RNA PCR (LOQ=50 copies/mL) assay will be used. It is noted that no testing outside of what is specified in this protocol, will be conducted without additional written informed consent.

LabCorps of America Monogram Phenosense GT will be performed in all patients at baseline and for all patients with confirmed virologic failure (two consecutive HIV RNA levels ≥400 copies/mL after suppression to <400 copies/mL for two consecutive measurements). Due to test reliability, HIV RNA must be ≥1000 copies/mL in order to obtain genotype. In patients with HIV RNA >500 but <1,000 copies/mL, testing may be unsuccessful but will be up to the discretion of the investigator. Genotypes will be utilized for use in clinical management.12subjects at their baseline and with at least 24 weeks exposure to darunavir and rilpivirine will have a sample of CSF for viral load, cell count and darunavir and rilpivirine concentration to be performed by LabCorps of America and by the University of California, San Diego, CA

Assessment of facial lipoatrophy, central adiposity, breast hypertrophy, dorsal fat pad ("buffalo hump"), multiple lipomas, and Cushingoid appearance without Cushing's disease will be performed by physician assessment and self-report at baseline, weeks 24, 48, and at premature discontinuation.

Patients who develop a study drug-related Grade 1 or 2 AE or clinical laboratory abnormality may elect to continue study medications. Patients who develop a study drug-related Grade 3 AE or clinical laboratory abnormality, with the exception of hyperglycemia, hypertriglyceridemia, hypercholesterolemia, or Grade 3 AST/ALT elevations, may interrupt the offending study medication(s) based on the discretion of the investigator. If only rilpivirine is determined to be the most likely most likely cause, darunavir/cobicistat may be continued for one additional week due to the long half-life of rilpivirine (~40 hours) to prevent functional monotherapy. Patients who develop a study drug-related Grade 4 AE or clinical laboratory abnormality, with the exception of hyperglycemia, hypertriglyceridemia, hypercholesterolemia, should interrupt all study medication, regardless of half-life. Upon resolution of the AE or clinical laboratory abnormality to within one grade level (not to exceed Grade 2) of the patient's baseline level, the patient may resume study drug dosing under the guidance of the investigator. Refer to Section 5 for more detailed information on toxicity management.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 RNA ≥ 5000 copies/mL by PCR
2. ≥ 18 years of age
3. Cognitive ability to understand and provide written informed consent and willingness to participate in and comply with the study protocol
4. Less than 7 days of prior ART with any licensed or investigational compound
5. Patient does not currently have or has not been treated for an active opportunistic infection (OI) consistent with CDC definition (Appendix C) within 30 days of screening
6. Vital signs, physical examination and laboratory results do not exhibit evidence of acute illness
7. A female is eligible to enter and participate in this study if she is of non child bearing potential or child bearing potential, has a negative serum pregnancy test at screen.

Exclusion Criteria

1. Patient with active AIDS-defining opportunistic infection or disease according to the 1993 CDC AIDS surveillance definition (Clinical Category C) in the 30 days prior to baseline and that, in the opinion of the investigator, would preclude the patient from participating in the study (See Appendix C).
2. Patient has none of the following darunavir-associated RAMs: V11I, V32I, L33F, I47V, I50V, I54L, I54M, T74P, L76V, I84V, L89V
3. Having documented genotypic evidence of NNRTI resistance at screening or from historical data available in the source documents, i.e. at least one of the NNRTI rams from the following list; K101E, K101P, E138A, E138G, E138K, E138R, E138Q, , V179L, Y181C, Y181I, Y181V, Y188L, H221Y, F227C, M230I, M230L, or the combination of the K103N and L100I.
4. History of active substance abuse, excluding cannabis, or psychiatric illness that, in the opinion of the investigator, would preclude compliance with protocol, dosing schedule and assessments.
5. Patient is either pregnant at time of screening evaluation or breast-feeding.
6. Patient, in the opinion of the investigator, is unlikely to be able to complete the 48-week dosing period and protocol evaluations and assessments or adhere to the study drug regimen.
7. Patient suffers from a serious medical condition, such as diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction, which in the opinion of the investigator would compromise the safety of the patient
8. Patient has malabsorption syndrome or other gastrointestinal dysfunction, which may interfere with drug absorption or render the patient unable to take oral medication.
9. Patient is undergoing interferon therapy for HCV or anticipates undergoing therapy during the course of this trial
10. HBV co-infection
11. Patient has any of the following laboratory results within 30 days prior to the first dose of study medication:

    * Hemoglobin concentration < 8.0 g/dL
    * Absolute neutrophil count < 750 cells/mm3
    * Platelet count <50,000 cells/ mm3
    * Aminotransferase (AST, ALT) >3 times ULN
    * Serum creatinine >1.5 times the Upper Limits of Normal (ULN)
12. Patients with severe hepatic impairment
13. Patient has required treatment with radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to entry, or has an anticipated need for these agents within the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA <50 copies/mL | up to weeks 48

SECONDARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA <400 copies/mL at each time point evaluated | At week 4, week 12, week 24, week 36, week 48
Number of weeks until HIV RNA <400 copies/mL and <50 copies/mL, respectively | At week 4, week 12, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Gathe, Jr., MD, Principal Investigator — Therapeutic Concepts, PA
Locations (2):
- United States (2):
  - Therapeutic Concepts, P.A., Houston, Texas
  - Therapeutic Concepts, PA, Houston, Texas